CLINICAL TRIAL: NCT06157970
Title: The Effect of Sphenopalatine Ganglion Block on Intraoperative Remifentanil Consumption and Postoperative Pain in Septorhinoplasty Surgery
Brief Title: Sphenopalatine Ganglion Block in Septorhinoplasty
Status: Completed | Type: Observational
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Suheda Akbulut, Principal Investigator, Istanbul Medeniyet University
Other Study IDs: MedeniyetUniverstySAkbulut001
Record Dates: First submitted 2023-11-08; First posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-12

CONDITIONS: Pain, Postoperative; Rhinoplasty
MeSH Terms: conditions — Pain, Postoperative | interventions — Sphenopalatine Ganglion Block

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Block Group: After intubation, the plastic part of the 18G angioket is placed transnasally into both nostrils in the supine position of the patients who will undergo sphenopalatine ganglion block, with the head in 15-20° extension and is advanced until it contacts the posterior mucosa. After contact, withdraw 1 mm and apply 0.5% bupivacaine 2 ml by dropping into the postnasal space within 1 minute.
  Interventions: Procedure: Sphenopalatine Ganglion Block
- Control Group: Group of patients who did not undergo sphenopalatine gangion block

INTERVENTIONS:
Procedure: Sphenopalatine Ganglion Block — For SPGB, the plastic part of the 16G angiogram is advanced transnasally into both nostrils, with the patient in the supine position and the head in 15-20° extension, until it contacts the posterior mucosa, and after contact, it is withdrawn 1 mm and 2 ml of 0.5% bupivacaine is dripped into the postnasal space within 1 minute. is applied.
  Groups: Block Group

SUMMARY:
Septorhinoplasty is a widely performed surgery that aims to correct both functional and aesthetic problems of the nose. Despite its expected clinical benefits, septorhinoplasty surgery causes postoperative pain, which affects the patient's functional recovery and satisfaction. Opioids, Non-steroidal anti-inflammatory drugs (NSAII), acetaminophen and local anesthetics are used in peroperative pain management in septorhinoplasty. Sphenopalatine ganglion block (SPGB), which has been recently described and has different application areas, is a regional analgesia technique that has been investigated for this purpose. Although there are studies on postoperative pain in septorhinoplasty surgeries, there are not enough studies on its effects on intraoperative pain.

This study may have positive effects on appropriate pain management, patient comfort and surgical outcomes as multimodal analgesia management in septorhinoplasty surgeries, and may make significant contributions to evidence-based practices.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing septorhinoplasty surgery
* Ages between 18-65
* ASA (American Society of Anesthesiologists) score I-II

Exclusion Criteria:

* Unavailable postoperative pain scores and analgesic use in the hospital registry system
* Local anesthetic drug allergy and toxicity
* Advanced organ failure
* Mental retardation

Patients who are pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who operated for septorhinoplasty
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-06-07 (Actual); Primary Completion 2023-08-21 (Actual); Study Completion 2023-08-21 (Actual)

PRIMARY OUTCOMES:
remifentanil consumption | 2 hours
  microgram

SECONDARY OUTCOMES:
Numerical Rating Scale | 15 minute, 30 minute, 1hour, 2 hour, 4 hour, 8 hour,16 hour, 24 hour
  Minimum values=1 and Maximum value=10. Highest values are worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Suheda Akbulut, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No